CLINICAL TRIAL: NCT01358942
Title: Observational, Epidemiological and Non Interventional Study Evaluating the Evolution of Lung Cancer Related Symptoms and Its Correlation With Disease Control Rate in Patients With Non-Small Cell Lung Cancer (NSCLC) Initiating First-line Treatment With Platinum Based Standard Chemotherapy.
Brief Title: An Observational Study of Lung Cancer Related Symptoms and Disease Control Rate in Patients With Non-Small Cell Lung Cancer Receiving First-Line Platinum-Based Chemotherapy With or Without Avastin (Bevacizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25493
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the evolution of lung cancer related symptoms and their correlation with the disease control rate (complete response, partial response and stable disease) in patients with non-small cell lung cancer initiating first-line treatment with standard platinum-based chemotherapy with or without Avastin (bevacizumab). Data will be collected from each patient at baseline and after 4-6 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed non-small cell lung cancer
* Initiating first-line treatment with standard platinum-based chemotherapy, with or without bevacizumab

Exclusion Criteria:

* Contraindications to the use of platinum-based chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients initiating treatment with platinum-based chemotherapy +/- bevacizumab
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in lung cancer related symptoms (LCSS questionnaire) | up to approximately 6 months (4-6 cycles of chemotherapy)
Correlation of lung cancer related symptoms and disease control rate (complete response, partial response, stable disease according to RECIST criteria) | approximately 2 years

SECONDARY OUTCOMES:
Frequency/severity of lung cancer related symptoms (LCSS questionnaire) | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Spain (27):
  - Vitoria-Gasteiz, Alava
  - Alcoy, Alicante
  - Alicante, Alicante
  - Elche, Alicante
  - Elda, Alicante
  - Maó, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Jerez de la Frontera, Cadiz
  - Castellon, Castellon
  - Donostia / San Sebastian, Guipuzcoa
  - Jaén, Jaen
  - Logroño, La Rioja
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Melilla, Malaga
  - Navarra, Navarre
  - Pamplona, Navarre
  - Tudela, Navarre
  - Pontevedra, Pontevedra
  - Oviedo, Principality of Asturias
  - Segovia, Segovia
  - Sagunto, Valencia
  - Valencia, Valencia
  - Xàtiva, Valencia
  - Bilbao, Vizcaya